CLINICAL TRIAL: NCT04686214
Title: The Effect of the Alterations in Body Temperature to Perioperative Bleeding in Adolescent Idiopathic Scoliosis Surgery
Brief Title: Body Temperature and Perioperative Bleeding in Adolescent Idiopathic Scoliosis Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nur Canbolat, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/145
Record Dates: First submitted 2020-12-18; First posted 2020-12-28 (Actual); Last update posted 2020-12-28 (Actual); Status verified 2020-12

CONDITIONS: Hypothermia; Anesthesia
MeSH Terms: conditions — Hypothermia | interventions — Heating

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental)
  Interventions: Procedure: heating
- control group (No Intervention)

INTERVENTIONS:
Procedure: heating — patients were aggressively warmed using multiple heating methods such as pressurized air heater and intravenous fluid heater
  Arms: study group

SUMMARY:
In this study, patient groups in which normothermia is preserved by using multiple active warming methods in the intraoperative period in AIS surgery, followed by a single compressed air blowing system and allowed mild to moderate hypothermia were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 12-18 who were evaluated as ASI by axial skeletal deformity, who would undergo elective deformity correction surgery, who did not have scoliosis due to a secondary cause, and whose data were allowed to be used by themselves and parents

Exclusion Criteria:

* Patients with body weight <35kg, morbid obesity (BMI> 40kg / m2), known allergy, known bleeding-coagulation disease, use of drugs that affect blood clotting parameters in the last week, presence of hepatic, renal, hematological, rheumatological disease, the patient's own or family with psychiatric disorders who could not cooperate

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
blood loss in the group of patients who are kept normothermic | surgery time (approximately 2 hours)
  to test that blood loss is reduced in the group of patients who are kept normothermic by applying aggressive multiple warming method compared to the patient group in which mild-moderate hypothermia was allowed by using a standard single heater in an operation that poses a high risk for bleeding and hypothermia, such as AIS deformity correction surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Faculty of Medicine, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gozubuyuk E, Aygun E, Basaran I, Canbolat N, Cavdaroglu B, Akgul T, Buget MI. Effects of Changes in Body Temperature on Perioperative Bleeding in Adolescent Idiopathic Scoliosis Surgery. Ther Hypothermia Temp Manag. 2022 Sep;12(3):146-154. doi: 10.1089/ther.2021.0016. Epub 2021 Oct 18. PMID 34665055